CLINICAL TRIAL: NCT00298688
Title: Phase II Study of Iressa in Relapsed and Refractory Small Cell Lung Cancer
Brief Title: A Study of IRESSA in Relapsed and Refractory Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0559
Record Dates: First submitted 2006-03-01; First posted 2006-03-03 (Estimated); Last update posted 2008-06-12 (Estimated); Status verified 2008-06

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Gefitinib

INTERVENTIONS:
Drug: Gefitinib

SUMMARY:
The purpose of this study is to determine the disease control rate at trial closure and after the first stage of the study in patients with relapsed or refractory SCLC and measurable disease treated with gefitinib

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Histologically confirmed, relapsed or refractory SCLCr
* Aged 18 or over and a life expectancy of more than 2 months

Exclusion Criteria:

* Any evidence of clinically active interstitial lung disease
* Other co-existing malignancies or malignancies diagnosed within the last 5 years, with the exception of basal cell carcinoma or cervical cancer in situ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56
Dates: Start 2004-09; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
To determine the disease control rate in these patients

SECONDARY OUTCOMES:
To determine the objective response rate at trail closure in these patients
To determine the time to progression-or-death in these patients
To determine overall survival in these patients

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Iressa Medical Science Director, MD, Study Director — AstraZeneca
Locations (3):
- Denmark (2):
  - Research Site, Copenhagen
  - Research Site, Herlev
- Research Site, Manchester, United Kingdom